CLINICAL TRIAL: NCT02342028
Title: Impact of Intermittent Hypoxia on the Number and Function of Regular T Cell in Patients With Obstructive Sleep Apnea
Brief Title: The Number and Function of Regular T Cell in Patients With Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Chou, Kun-Ta, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 2015-01-005AC
Record Dates: First submitted 2015-01-12; First posted 2015-01-19 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Sleep Apnea Syndromes
Keywords: sleep apnea; intermittent hypoxia; regulatory T cell; autoimmunity
MeSH Terms: conditions — Sleep Apnea Syndromes; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — the whole blood of enrollees
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OSA: The study group enrolled patients with OSA, fulfilling the following requirements
  1. 20~60 years ago, female or males
  2. Agree participate the study and sign informed consent
  3. Has not received any treatment for OSA
  4. No obvious comorbidities (including autoimmune diseases)
  5. No history of sarcoidosis and tuberculosis
  6. No use of steroid and immunosuppressant
  Interventions: Biological: OSA
- Control: The control group enrolled age-, gender- and BMI-matched individuals without OSA, fulfilling the following requirements
  1. 20~60 years ago, female or males
  2. Agree participate the study and sign informed consent
  3. No obvious comorbidities (including autoimmune diseases)
  4. No history of sarcoidosis and tuberculosis
  5. No use of steroid and immunosuppressant

INTERVENTIONS:
Biological: OSA — This study aims to compare the difference in the number and function of regulatory T cells between OSA patients and controls. The investigators will draw peripheral venous blood samples from both groups and measure the number and function of their regulatory T cells. However, some, NOT ALL, of OSA patients may receive continuous positive airway pressure (CPAP) treatment-the standard therapy for severe-to-moderate OSA. Use of CPAP is based on physician's suggestion and patients' decision, but not for this study. The devices are provided by patients themselves and its type/brand is not limited or prespecified. For those with CPAP therapy, their blood sample will be re-collected 26 weeks later to repeat measurement for subgroup analysis.
  Groups: OSA

SUMMARY:
To compare the number and function of regular T cell of patients with obstructive sleep apnea (OSA) versus that of age-, gender- and BMI (body mass index)-matched controls

DETAILED DESCRIPTION:
Patients with obstructive sleep apnea (OSA) experience intermittent hypoxemia and arousal during sleep due to recurrent collapse of upper airway. Epidemiologic evidence showed they were at higher risk for autoimmune diseases. The regular T cell (Treg) has a crucial role in controlling autoimmunity. In this study, 40 OSA patients and 40 age-, gender- and BMI-matched controls will be recruited. Peripheral venous blood of the participants is drawn for numeration of CD4+CD25+FoxP3+ regular T cells by flow cytometry. As well, the CD4+CD25+ regular T cells are enriched by MACS and tested for their suppressive functions on proliferation assays. Th12+ CD4+ cells are also measured.

ELIGIBILITY:
Inclusion Criteria:

1. OSA patients diagnosed with a polysomnography
2. Agree to participate the study and sign informed consent

Exclusion Criteria:

1. Do not agree to participate the study and sign informed consent
2. Has received any treatment or OSA
3. With major comorbidities (such as a diabetes, heart disease, lung diseases, renal diseases, autoimmune diseases, but hypertension excluded)
4. History of sarcoidosis and tuberculosis
5. On treatment of steroid and immunosuppressant

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: OSA patients free of other specific conditions affecting immunity are enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The number and function of regular T cells in peripheral venous blood | 0-26 week

SECONDARY OUTCOMES:
The number of Th12+ CD4+ cells | 0-26 week

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ta Chou, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Chest department, Taipei Veteran General Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Chou KT, Liu CC, Hsu HS, Chang SC, Chen YM, Perng DW, Hsu YT, Lee YC, Hung SC. Nocturnal stem cell mobilization in patients with obstructive sleep apnoea: a pilot study. Eur J Clin Invest. 2014 Dec;44(12):1189-96. doi: 10.1111/eci.12353. PMID 25331065
- [Background] Kotsianidis I, Nakou E, Bouchliou I, Tzouvelekis A, Spanoudakis E, Steiropoulos P, Sotiriou I, Aidinis V, Margaritis D, Tsatalas C, Bouros D. Global impairment of CD4+CD25+FOXP3+ regulatory T cells in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2009 Jun 15;179(12):1121-30. doi: 10.1164/rccm.200812-1936OC. Epub 2009 Apr 2. PMID 19342412